CLINICAL TRIAL: NCT04782219
Title: Reliability and Validity of the Turkish Version of Patient-Reported Outcomes Measurement Information System-29 in Individuals With Musculoskeletal Diseases
Brief Title: Validity of Turkish Version of PROMIS-29 Measure
Status: Completed | Type: Observational
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Burcu Özdemir Kocabey, MSc, PhD(c), Bahçeşehir University
Other Study IDs: AcibademH
Record Dates: First submitted 2021-02-28; First posted 2021-03-04 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Musculoskeletal Diseases
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will be carried out on 100 patients with chronic musculoskeletal disorders who applied to Acıbadem Maslak Hospital Orthopedics and Traumatology Department. Demographic information (age, education level, occupation, marital status) will be obtained from the patients, they will be asked whether they have a chronic musculoskeletal disease diagnosed by the doctor, and they will be asked to fill in the PROMIS 29 and SF-36 v2 questionnaires.

The PROMIS 29 questionnaire contains 4 questions from each of the seven contents of PROMIS (physical function, depression, anxiety, fatigue, sleep disorder, participation in social activities and pain interaction) and 1 question from the intensity of pain. Each item has 5 answer options (from 1 to 5), only pain intensity has 11 answer options (from 0 to 10). From the sum of the answers to each question in the domain, the total raw score for each domain is calculated, resulting in seven domain scores, each between 4 and 20. SF-36 is the most widely used scale to assess general health status, and 36 items question 8 content (physical function, physical role, pain, general health, social function, energy / fitness, social function, emotional role, mental health). The Turkish translation of the PROMIS 29 questionnaire is presented in ANNEX-2.

The translation of the PROMIS 29 questionnaire into Turkish was made by Northwestern University according to the FACIT translation method. Its Turkish translation was obtained from Northwestern University by signing a license agreement for use in scientific research.

Participants will first be asked to sign the informed consent form electronically. PROMIS 29 and SF-36 v2 forms will be sent to the volunteers via e-mail and will be asked to respond via an internet-based questionnaire platform.

The external validity of the PROMIS 29 questionnaire will be evaluated by its correlation with the SF-36 v2, a similar general health profile questionnaire.

To evaluate inter-rater test-retest reliability, both scales will be filled in by patients a second time between 7-14 days.

ELIGIBILITY:
Inclusion Criteria:

* Being over the age of 18,
* To be able to read and speak Turkish,
* To have a chronic musculoskeletal disease
* volunteering to participate in the study

Exclusion Criteria:

* To have serious medical conditions or complications (such as vision or hearing impairments) that may affect the participant's ability to respond to study questionnaires

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons who applied to the Acibadem Maslak Hospital Orthopedics and Traumatology department and were diagnosed with a chronic musculoskeletal disease by orthopedists will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-03-20 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Patient Reported Outcome Measures Information System-29 (PROMIS-29) | It will be filled for the second time between 7-14 days.
  The PROMIS 29 questionnaire contains 4 questions from each of seven PROMIS contents (physical function, depression, anxiety, fatigue, sleep disorder, participation in social activities and pain interaction) and 1 question from the intensity of pain. Each item has 5 answer options (from 1 to 5), only pain intensity has 11 answer options (from 0 to 10). From the sum of the answers to each question in the domain, the total raw score for each domain is calculated, resulting in seven domain scores, each between 4 and 20.
Short Form-36 (SF-36) | It will be filled for the second time between 7-14 days.
  SF-36 is the most widely used scale to assess general health status, and 36 items question 8 content (physical function, physical role, pain, general health, social function, energy / fitness, social function, emotional role, mental health)

CONTACTS AND LOCATIONS:
Overall Officials: Göksel Dikmen, Assoc. Prof., Principal Investigator — Acibadem University
Locations (1):
- Maslak Acıbadem Hospital, Istanbul, Turkey (Türkiye)